CLINICAL TRIAL: NCT01442519
Title: Sequential Bacillus Calmette-Guérin and Electromotive Mitomycin-C Versus Bacillus Calmette-Guérin Alone for High Risk Superficial Bladder Cancer: a Prospective Randomised Study
Brief Title: Sequential Bacillus Calmette-Guérin (BCG) and Electromotive Mitomycin-C Versus Bacillus Calmette-Guérin (BCG) Alone for High Risk Superficial Bladder Cancer
Acronym: BCG/EMDA-MMC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Savino M. Di Stasi, Professor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTV-119-1993
Record Dates: First submitted 2011-07-29; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Bladder Cancer
Keywords: non-muscle invasive urothelial bladder cancer; intravesical therapy; BCG; mitomycin; electromotive drug administration; Bladder Cancer Stage 0, Without Cancer in Situ
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine; BCG Connaught; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravesical BCG alone (Active Comparator)
  Interventions: Biological: bacillus Calmette-Guerin
- Intravesical sequential BCG and EMDA MMC (Experimental)
  Interventions: Drug: electromotive mitomycin

INTERVENTIONS:
Biological: bacillus Calmette-Guerin — The BCG instillation consisted of 81 mg wet weight (10•2±9•0_108 colony-forming units) BCG Connaught substrain (ImmuCyst®, Alfa Wassermann SpA, Bologna, Italy). Lyophilised (ie, freeze-dried) BCG is suspended in 50 mL bacteriostatic-free solution of 0•9% sodium chloride. After draining of the bladder, the suspension is infused intravesically through a Foley catheter. The solution is retained in the bladder for 120 min, followed by emptying of the bladder and removal of the catheter. The BCG-alone group is assigned one course of intravesical treatment per week for 6 weeks. Patients in the BCG-alone group who are disease-free 3 months after treatment are scheduled to receive monthly infusions of BCG for 10 months
  Other Names: IMMUCYST, Alpha Wassermann, Bologna, Italy
  Arms: Intravesical BCG alone
Drug: electromotive mitomycin — BCG instillation of 81 mg BCG Connaught-substrain, suspended in 50 mL bacteriostatic-free saline solution, retained for 120 min. Electromotive instillation: 40 mg mitomycin in 100 mL water infused intravesically and retained in the bladder for 30 min, while 20 mA for 30 min pulsed electric current is given externally. Patients assigned sequential BCG and EMDA MMC are assigned 1 course of treatment/week for 9 weeks: one cycle consisted of two BCG infusions and one mitomycin infusion (three cycles in total). Patients in the BCG-and-mitomycin group who are disease-free 3 months after treatment are scheduled to receive one infusion a month for 9 months: three cycles of mitomycin, mitomycin, and BCG (ie, six infusions of MMC and three of BCG).
  Other Names: IMMUCYST, Alpha Wassermann, Bologna, Italy; MITOMYCIN C 40 mg, Kyowa Italiana Farmaceutici
  Arms: Intravesical sequential BCG and EMDA MMC

SUMMARY:
Intravesical treatment for superficial bladder cancer has been used for the past 4-5 decades. Intravesical chemotherapy is beneficial in terms of recurrence and time to recurrence in grade 1-2 stage Ta tumours, usually non-invasive. Intravesical chemotherapy has negligible effect on disease progression in high-risk superficial bladder cancer-ie, grade 3, stage T1, and carcinoma in situ. However, BCG as induction and maintenance treatment effectively delays progression. Electromotive mitomycin increases tissue uptake compared with that of passive diffusion. Electromotive mitomycin has emerged as an alternative or complementary treatment to BCG. The rationale for combining anticancer drugs is based on the need to increase efficacy and reduce emergence of resistant malignant cells. This approach is not frequently applied to use of intravesical agents for treatment of superficial bladder cancer, for which immunotherapeutic BCG and chemotherapeutic mitomycin seem to be a potentially effective combination. Studies have addressed concurrent use of mitomycin and BCG, and assigned two roles to mitomycin: antitumor action and tissue-scarifying (ie, surface-modifying) effect that enables BCG to attach more efficiently to the urothelium. The investigators therefore aimed to assess whether induction of inflammation by use of BCG before mitomycin treatment makes the bladder mucosa more permeable and thus enables mitomycin to reach the target more easily. This randomised trial to compare the efficacy of sequential BCG and electromotive mitomycin with that of the current standard of BCG alone for patients with high-risk superficial bladder cancer.

After transurethral resection and multiple biopsies patients with stage pT1 bladder cancer are randomly assigned to: 81 mg BCG infused over 120 min once a week for 6 weeks; or to 81 mg BCG infused over 120 min once a week for 2 weeks, followed by 40 mg electromotive mitomycin (intravesical electric current 20 mA for 30 min) once a week as one cycle for three cycles (n=107). Complete responders underwent maintenance treatment: those assigned BCG alone had one infusion of 81 mg BCG once a month for 10 months, and those assigned BCG and mitomycin had 40 mg electromotive mitomycin once a month for 2 months, followed by 81 mg BCG once a month as one cycle for three cycles. The primary endpoint was disease-free interval; secondary endpoints were time to progression; overall survival; and disease-specific survival. Analyses were intention to treat.

DETAILED DESCRIPTION:
All patients with histologically proven stage pT1 urothelial carcinoma of the bladder, whether papillary or solid, are regarded as being at high risk for tumour recurrence and at moderate to high risk for progression because of: multifocal pT1, primary or recurrent, grade 2 transitional-cell carcinoma; primary or recurrent pT1, multifocal or solitary, grade 3 transitional-cell carcinoma; or pT1 with carcinoma in situ. Inclusion criteria are: age 18 years or older; adequate bone-marrow reserve; normal renal function; normal liver function; and Karnofsky performance status between 50 and 100. Exclusion criteria are: previous treatment with BCG or electromotive mitomycin; treatment with any other intravesical cytostatic agent within the past 6 months; concomitant urothelial tumours of the upper urinary tract; previous muscle-invasive (ie, stage T2 or higher) transitional-cell carcinoma of the bladder; bladder capacity less than 2 L; untreated urinary-tract infection; severe systemic infection (ie, sepsis); urethral strictures that would prevent endoscopic procedures and repeated catheterisation; disease of upper urinary tract (eg, vesicoureteral reflux or urinary-tract stones) that would make multiple transurethral procedures a risk; previous radiotherapy to the pelvis; other concurrent chemotherapy; treatment with radiotherapy-response or biological-response modifiers; history of tuberculosis; other malignant diseases within 5 years of trial registration (except for basal-cell carcinoma); pregnancy or nursing; and psychological, familial, sociological, or geographical factors that would preclude study participation.

Study design The institutional review boards of every participating centre approved the study design. Every patient enrolled signed an informed-consent form approved by the institutional review boards. All patients underwent: urinary cytology of the bladder and upper urinary tract; random cold-cup biopsies of the bladder and prostatic urethra-ie, sampling of seemingly healthy urothelium and of suspicious areas; and complete transurethral resection of all bladder tumour visible on endoscopy, ensuring muscle is included in resected samples. Patients with positive or suspect cytology, carcinoma in situ, multifocal tumours, or grade 3 tumours underwent restaging transurethral resection 4-5 weeks later. All clinical assessors are adequately trained in the above procedures, and no methods are used to enhance the quality of measurements. All biopsy samples of tumour and bladder are reviewed by a pathologist for stage and grade. Tumour stage is classified according to the 1997 TNM classification of the International Union Against Cancer, and tumour grade is defined in accordance with the 1973 WHO classification. Patients are randomised within 10 days of the first or restaging transurethral resection. Randomisation and data collection are done by use of a central computer. Patients are allocated to BCG alone or to BCG and electromotive mitomycin by use stratified, blocked randomisation cross 14 strata as a result of four factors: primary versus recurrent tumours; multifocal versus unifocal tumours; grade 3 versus grade 2 tumours; and presence versus absence of carcinoma in situ. MV generated and coordinated the randomisation process. This study is not blinded because of differences in treatment schedules and drug appearance.

Treatment schedules All patients are scheduled to receive their allocated intervention about 3 weeks after transurethral resection and multiple, random biopsy sampling. The BCG instillation consisted of 81 mg wet weight BCG Connaught substrain (ImmuCyst®, Alfa Wassermann SpA, Bologna, Italy). Lyophilised (ie, freeze-dried) BCG is suspended in 50 mL bacteriostatic-free solution of 0·9% sodium chloride. After draining of the bladder, the suspension is infused intravesically through a Foley catheter. The solution is retained in the bladder for 120 min, followed by emptying of the bladder and removal of the catheter. Patients randomly allocated to BCG and mitomycin, are placed on fluid restriction and 2 g ingested sodium bicarbonate the night before treatment, the morning of treatment, and 2 h before treatment with mitomycin. A Foley catheter is inserted and postvoid residual volume is reduced to less than 10mL. 40 mg mitomycin (Mitomycin, Kyowa Italiana Farmaceutici, Srl, Milan, Italy) dissolved in 100 mL water is infused intravesically through the Foley catheter by gravity and retained in the bladder for 30 min, while 40-60 mA per s to a maximum of 20 mA or 30 min pulsed electric current is given externally.13 Two dispersive cathode electrodes are placed on lower abdominal skin that had been degreased with alcohol and a 2-5-mm layer of conductive gel applied. The bladder is then emptied and the catheter removed. The BCG-alone group is assigned one course of intravesical treatment per week for 6 weeks; patients assigned sequential BCG and electromotive mitomycin are assigned one course of treatment per week for 9 weeks, for whom one cycle consisted of two BCG infusions and one mitomycin infusion (three cycles in total). Patients in the BCG-alone group who are disease-free 3 months after treatment are scheduled to receive monthly infusions of BCG for 10 months. Patients in the BCG-and-mitomycin group who are disease-free 3 months after treatment are scheduled to receive one infusion a month for 9 months: three cycles of mitomycin, mitomycin, and BCG (ie, six infusions of mitomycin and three infusions of BCG.

Maintenance treatment for both groups is given to the same dose and methods of infusion as initial allocated treatment.

Role of the funding source The sponsor of the study has no role in study design; in the collection, analysis, or interpretation of data; or in the writing of the report.

ELIGIBILITY:
Inclusion Criteria:

* adequate bone-marrow reserve (ie, white-blood-cell count ≥4000 x106 cells/L and platelet count ≥120 x 109/L)
* normal renal function (ie, serum creatinine ≤123•76 μmol/L)
* normal liver function (ie, serum glutamic-oxaloacetic transaminase ≤42 U/L, serum glutamic-pyruvic transaminase ≤48 U/L, and total bilirubin ≤22•23 μmol/L)
* Karnofsky performance status between 50 and 100.

Exclusion Criteria:

* previous treatment with BCG or electromotive mitomycin
* treatment with any other intravesical cytostatic agent within the past 6 months
* concomitant urothelial tumours of the upper urinary tract;
* previous muscle-invasive (ie, stage T2 or higher) transitional-cell - carcinoma of the bladder
* bladder capacity less than 2 L
* untreated urinary-tract infection
* severe systemic infection (ie, sepsis)
* urethral strictures that would prevent endoscopic procedures and repeated catheterisation
* disease of upper urinary tract (eg, vesicoureteral reflux or urinary-tract stones) that would make multiple transurethral procedures a risk
* previous radiotherapy to the pelvis
* other concurrent chemotherapy
* treatment with radiotherapy-response or biological-response modifiers;
* history of tuberculosis
* other malignant diseases within 5 years of trial registration (except for basal-cell carcinoma)
* pregnancy or nursing
* psychological, familial, sociological, or geographical factors that would preclude study participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 1994-01; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Disease-free interval | From date of randomization until the date of first documented recurrence, assessed up to 120 months
  The primary endpoint is disease-free interval for patients without carcinoma in situ and for patients with carcinoma in situ who are disease-free after treatment-ie, time from randomisation to first cystoscopy noting recurrence. Patients with carcinoma in situ who did not have complete response after 3 months of treatment are regarded as having recurrence with no follow-up.

SECONDARY OUTCOMES:
Time to progression | From date of randomization until the date of documented progression, assessed up to 120 months.
  Time to progression is defined as time from randomisation until the onset of muscle-invasive disease as recorded by pathological assessment of transurethral-resection samples or biopsy samples. Patients without recurrence or progression are censored at the last cystoscopy, and those lost to follow-up are censored at the last known day of survival.
Overall survival | From date of randomization until the date of death for any cause, assessed up to 120 months.
  Overall survival is defined as time from randomisation until death from any cause. Patients without recurrence or progression are censored at the last cystoscopy, and those lost to follow-up are censored at the last known day of survival.
Disease-specific survival | From date of randomization until the date of death for bladder cancer, assessed up to 120 months.
  Disease-specific survival as time from randomisation until death from bladder cancer. Patients without recurrence or progression are censored at the last cystoscopy, and those lost to follow-up are censored at the last known day of survival.

CONTACTS AND LOCATIONS:
Overall Officials: Savino M Di Stasi, MD, PhD, Principal Investigator — Tor Vergata University, Rome, Italy
Locations (1):
- Dept. of Surgery/Urology, Tor Vergata University, Rome, RM, Italy

REFERENCES:
- [Result] Di Stasi SM, Giannantoni A, Giurioli A, Valenti M, Zampa G, Storti L, Attisani F, De Carolis A, Capelli G, Vespasiani G, Stephen RL. Sequential BCG and electromotive mitomycin versus BCG alone for high-risk superficial bladder cancer: a randomised controlled trial. Lancet Oncol. 2006 Jan;7(1):43-51. doi: 10.1016/S1470-2045(05)70472-1. PMID 16389183